CLINICAL TRIAL: NCT00132743
Title: Claudication: Exercise Versus Endoluminal Revascularization (CLEVER)
Acronym: CLEVER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Joselyn Cerezo, MD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Joselyn Cerezo, MD, Clinical Trials Project Manager, Rhode Island Hospital
Organization: Rhode Island Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 224; U01HL081656 (NIH); U01HL077221 (NIH)
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Cardiovascular Diseases; Peripheral Vascular Diseases; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Peripheral Vascular Diseases; Atherosclerosis | interventions — Stents; Cilostazol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Optimal Medical Care
  Interventions: Behavioral: Supervised Exercise Therapy; Drug: Cilostazol
- 2 (Active Comparator): Optimal Medical Care and Supervised Exercise
  Interventions: Device: Stent; Drug: Cilostazol
- 3 (Active Comparator): Optimal Medical Care and Stent
  Interventions: Device: Stent; Behavioral: Supervised Exercise Therapy

INTERVENTIONS:
Device: Stent — Stent
  Arms: 2; 3
Behavioral: Supervised Exercise Therapy — Supervised exercise therapy, three times per week
  Arms: 1; 3
Drug: Cilostazol — Cilostazol, 100 mg twice a day
  Arms: 1; 2

SUMMARY:
The purpose of this study is to compare the effectiveness of aortic stent surgery versus exercise therapy in individuals with aortoiliac insufficiency.

DETAILED DESCRIPTION:
BACKGROUND:

Peripheral arterial disease (PAD) is a major source of morbidity and mortality, particularly in older individuals. Despite its high prevalence, clinicians often fail to diagnose PAD, particularly in patients who do not have classic claudication symptoms. Even in those individuals with documented PAD, cardiac risk factors are not often aggressively treated, and only a minority of patients receive pharmacologic therapy with cilostazol. Although there is a growing body of literature demonstrating the value of exercise rehabilitation in individuals with peripheral vascular disease and claudication, exercise rehabilitation is not often prescribed as supervised exercise rehabilitation for claudication, is not reimbursed by Medicare, and is rarely covered by private insurance. Therefore, few individuals with PAD and intermittent claudication have access to supervised exercise rehabilitation.

The use of surgical intervention and stent placement to improve blood flow in patients who do not have ischemic pain at rest or limb-threatening ischemia (Fontaine class III or IV) remains controversial. There is data suggesting that patients with intermittent claudication who have had revascularization with stents have improved exercise capacity and walking times. However, the patients in the various studies often differ substantially in their clinical characteristics, and a variety of techniques were employed, including balloon angioplasty and stents, which makes it difficult to come to a definitive conclusion about the relative efficacy of stenting to improve functional performance. Additionally, to our knowledge, the combination of stent revascularization with supervised exercise rehabilitation has not been studied.

DESIGN NARRATIVE:

The broad objective of the study is to optimize physical functioning, increase activity levels, and reduce cardiovascular disease risk in older individuals with PAD. The specific aim of the trial is to test the primary hypothesis that aortoiliac stenting/pharmacotherapy improves maximum walking duration (MWD) better than supervised exercise rehabilitation/exercise maintenance/pharmacotherapy for those with aortoiliac artery obstruction at 6 months. Other aims are to compare these two treatment groups with two other treatment groups, optimal medical care/pharmacotherapy and combined stent plus supervised exercise rehabilitation, at 6 months, and to compare all 4 groups with regard to the following variables: MWD change score at 18 months, changes in free-living daily activity levels, patient-perceived quality of life (QoL), and cost-effectiveness. The study also will perform exploratory analyses of demographic and biochemical risk factors for atherosclerosis, including body mass index (BMI), blood pressure, lipid profile, hemoglobin Alc (HgbAlc), fibrinogen, and C-reactive protein. An estimated 252 patients (at up to 30 study sites) with aortoiliac insufficiency and intermittent claudication will be randomly divided into four groups: optimal medical care/pharmacotherapy, supervised exercise rehabilitation/maintenance/pharmacotherapy, stent/pharmacotherapy, and stent/supervised exercise rehabilitation/pharmacotherapy. Recruitment will be performed over 28 months and patients will be followed for 18 months; the total study duration will be 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject has symptoms suggestive of intermittent claudication, such as exercise-induced pain, cramps, fatigue, or other equivalent discomfort, involving large muscle groups of the leg(s) (calf, thigh, buttocks), relieved by rest
* Claudication score consistent with "Rose", "atypical", or "noncalf" claudication by San Diego Claudication Questionnaire
* Positive noninvasive evaluation for significant aortoiliac PAD on the most symptomatic side(s) (bilaterally if symptoms are equal):

  * Contrast Arteriography: Contrast arteriogram showing at least 50% stenosis in the aorta, common iliac artery, or external iliac artery, OR
  * CTA or MRA: Ankle-brachial index less than or equal to 0.9 (or abnormal ankle PVR waveform at ankle if arteries are incompressible*) with at least 60% stenosis in the aorta, common iliac artery, external iliac artery, accompanied by a biphasic or monophasic Doppler wave form at the common femoral artery (loss of early diastolic flow reversal or loss of forward flow during diastole), OR
  * Duplex Ultrasound: Ankle-brachial index less than or equal to 0.9 (or abnormal ankle PVR waveform at ankle if arteries are incompressible*) with occlusion or focal doubling of peak systolic velocity in the aorta, common iliac artery, or external iliac artery, accompanied by a biphasic or monophasic Doppler wave form at the common femoral artery (loss of early diastolic flow reversal or loss of forward flow during diastole), OR
  * Vascular Noninvasive Physiologic Tests: Ankle-brachial index less than or equal to 0.9 (or abnormal ankle PVR waveform at ankle if arteries are incompressible*) with resting thigh-brachial index (thigh-BI) less than 1.1, and common femoral artery Doppler systolic acceleration time greater than 140 msec [these tests may be ordered for study screening].

    * Abnormal PVR waveform must lack augmentation at the ankle, have a delayed, rounded systolic peak, and straight or convex downslope, and must be reviewed by the core lab.

Note: MRA/CTA, and contrast arteriogram images images must be submitted to the Clinical Coordinating Center and Doppler waveform tracings to the Noninvasive Test Committee for over read pre- or post-randomization

* Highest ankle pressure reduced by at least 25 mm Hg after exercise compared to resting pressure (or loss of previously present Doppler signal for both the posterior tibial and anterior tibial arteries immediately after exercise if arteries were incompressible) Note: The highest ankle pressure result is determined by using the higher result of either the dorsalis pedis or posterior tibial artery measurement.
* Subject has moderate to severe claudication symptoms, defined as less than 11 minutes MWD at baseline (initial) Gardner treadmill test

Exclusion Criteria:

* Presence of critical limb ischemia (Rutherford Grade II or III59 PAD, defined as pain at rest, ischemic ulceration, gangrene) or acute limb ischemia (pain, pallor, pulselessness, paresthesias, paralysis) in either leg
* Common femoral artery (CFA) occlusion or greater than or equal to 50% stenosis by angiography, MRA, CTA, or duplex ultrasound or doubling of systolic velocity in the ipsilateral common femoral artery by duplex ultrasound, or 50% diameter stenosis by visual estimate in the CFA by angiography, MRA, or CTA, (inadequate outflow for iliac stent intervention), if available pre-randomization
* Known total aortoiliac occlusion from the renal arteries to the inguinal ligaments (all other occlusions, including aortic occlusion, ARE eligible)
* Participant has bilateral claudication symptoms and the limb that is more symptomatic does not show evidence of aortoiliac insufficiency as described in inclusion criterion number 5
* Participant has bilateral claudication symptoms, but both limbs are equally symptomatic and one side does not show evidence of aortoiliac insufficiency as described in inclusion criterion number 5
* Subject meets the following exclusions based upon modified American College of Sports Medicine criteria for exercise training:

  i. Ambulation limited by co-morbid condition other than claudication, for example:1. severe coronary artery disease; 2. angina pectoris; 3. chronic lung disease;4. neurological disorder such as hemiparesis;5. arthritis, or other musculoskeletal conditions including amputation ii. Poorly-controlled hypertension (SBP greater than 180 mm Hg) iii.Poorly-controlled diabetes mellitus iv. Other active significant medical problems such as cancer, known chronic renal disease (serum creatinine greater than 2.0 mg/dl within 60 days or renal replacement therapy), known chronic liver disease or anemia, active substance abuse, or known history of dementia
* Contraindication to exercise testing according to AHA/ACC guideline, specifically: Acute myocardial infarction (within 3-5 days), unstable angina, uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise, active endocarditis, symptomatic severe aortic stenosis, acute pulmonary embolus or pulmonary infarction, acute noncardiac disorder that may affect exercise performance or be aggravated by exercise such as infection, thyrotoxicosis, acute myocarditis or pericarditis, known physical disability that would preclude safe and adequate test performance, known thrombosis of the lower extremity, known left main coronary stenosis or its equivalent, moderate stenotic valvular heart disease, electrolyte abnormalities, known pulmonary hypertension, tachyarrhythmias or bradyarrhythmias, hypertrophic cardiomyopathy, mental impairment leading to inability to cooperate, or high degree atrioventricular block
* Arterial insufficiency of target lesion due to restenosis of an angioplasty/stent or bypass is not eligible
* Recent (less than 3 months) infrainguinal revascularization (surgery or endovascular intervention)
* Recent major surgery in the last 3 months
* Abdominal aortic aneurysm greater than 4 cm or iliac artery aneurysm greater than 1.5 cm is present
* Patients who are pregnant, planning to become pregnant, or lactating
* Unwilling or unable to attend regular (3 times a week) supervised exercise sessions. (Please review this commitment carefully with each prospective participant.)
* Weight greater than 350 lbs or 159 kg (may exceed treadmill and angiography table limits)
* Inability to understand and sign informed consent forms due to cognitive or language barriers (interpreter permitted)
* Absolute contraindication to iodinated contrast due to prior near-fatal anaphylactoid reaction (laryngospasm, bronchospasm, cardiorespiratory collapse, or equivalent) and which would preclude patient from participation in angiographic procedures
* Allergy to stainless steel or nitinol
* Allergy or other intolerance to cilostazol (bleeding history) or history of congestive heart failure [if ejection fraction is shown to be greater than or equal to 50% patient may be enrolled]
* Nonatherosclerotic cause of PAD (fibromuscular dysplasia, dissection, trauma, etc)
* Inability to walk on a treadmill without grade at a speed of at least 2 mph for at least 2 minutes on the first treadmill test
* ST-segment depression greater than 1 mm in any of the standard 12 ECG leads or sustained (greater than 30 seconds) arrhythmia other than tachycardia or occasional premature atrial or ventricular contractions during exercise testing
* Post-exercise systolic blood pressure within the first five minutes after eligibility treadmill test lower than pre-exercise systolic blood pressure
* A peak heart rate greater than 80% of maximum (calculated by subtracting age from 220) while reporting "onset" of claudication symptoms (level 3 or 4) during the second baseline examination
* Repeat treadmill test shows a MWD result that is greater than 25% different than the subject's initial Gardner treadmill test result. Current active involvement in a supervised exercise program (e.g., with a trainer, exercise protocol, and goals, such as in cardiac or pulmonary rehabilitation) for more than 2 weeks within the prior 6 weeks.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2007-02; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
MWD change score | Measured at 6 months
  Aortoiliac revascularization with stent (ST) combined with optimal medical care (OMC) improves maximum walking duration (MWD) compared to optimal medical care alone in patients with claudication and peripheral arterial disease (PAD) who are amenable to peripheral stenting
MWD change score | Measured at 6 months
  Regular supervised exercise (SE) combined with optimal medical care (OMC) improves maximum walking duration compared to optimal medical care along in patients with claudication and PAD who are amenable to peripheral stenting.
MWD change score | Measured at 6 months
  Aortoiliac revascularization with stent (ST) combined with optimal medical care improves maximum walking duration compared to supervised exercise (SE) combined with optimal medical care in patients with claudication and PAD who are amenable to peripheral stenting.

SECONDARY OUTCOMES:
MWD change score | Measured at 18 months
  To evaluate the mid-term durability of any treatment effect by performing pair-wise comparison of change in MWD between baseline and 18 month time points among all three treatment groups of primary interest.
Free-living daily activity | Measured at 6 and 18 months
  To assess a treatment effect on free-living daily activity levels of any treatment group, comparing baseline electronic step monitors values with those obtained at both follow up intervals (6 and 18 months)
Quality of Life | Measured at 6 and 18 months
  To examine treatment effects on patient-perceived health-related quality of life (physical function) between all groups at 6 and 18 months
Cost-effectiveness | Measured at 18 months
  To Examine inpatient and outpatient costs associated with the three treatment strategies, and to evaluate the relative cost-benefit by calculating incremental cost-effectiveness and cost effectiveness acceptability curves using health utility change in the denominator.
Cardiovascular risk factors | Measured at baseline, 6 months, and 18 months
  To evaluate the impact of cardiovascular disease risk factors by comparing these values at baseline, 6 months, and 18 months.
Interaction effect | Measured at 18 months
  To evaluate the interaction effect, if any, of gender or race on improvements in MWD, improvement in free-living daily activities, and quality-of-life.
Major adverse peripheral events | Measured from randomization to 18 months
  To track major adverse peripheral events (MAPEs) associated with aortoiliac stenting and femoropopliteal endovascular intervention.
Major complication | Measured from randomization to 18 months
  Rate of major complication defined as any occurrence of death, myocardial infarction, amputation of the target limb (limb treated in this study), or occurrence of critical limb ischemia or repeat target limb revascularization (TLiR).

CONTACTS AND LOCATIONS:
Overall Officials: Don Cutlip, MD, Principal Investigator — Brigham and Women's Hospital; Timothy Murphy, MD, Principal Investigator — Rhode Island Hospital
Locations (27):
- United States (26):
  - VA Loma Linda, Loma Linda, California
  - St. Joseph Hospital, Orange, California
  - VA Palo Alto Health Care Systems, Palo Alto, California
  - UC Davis, Sacramento, California
  - Vasek Polak Research Program, Torrance, California
  - Baptist Cardiac and Vascular Institute, Miami, Florida
  - Aiyan Diabetes Center, Evans, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The Iowa Clinic, Des Moines, Iowa
  - Rapides Regional Medical Center, Alexandria, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins, Baltimore, Maryland
  - VA Ann Arbor, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Abbott Northwestern Vascular Center, Minneapolis, Minnesota
  - Stony Brook, Stony Brook, New York
  - Asheville Cardiology, Asheville, North Carolina
  - Forsyth-Salem Surgical, Winston-Salem, North Carolina
  - Vascular Endovascular Specialists of Ohio, Mansfield, Ohio
  - Jobst Vascular, Toledo, Ohio
  - Oregon Health Science University (DOTTER), Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Providence Medical Research, Spokane, Washington
  - Charleston Area Medical Center, Charleston, West Virginia
- Capital Health, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Bronas UG, Hirsch AT, Murphy T, Badenhop D, Collins TC, Ehrman JK, Ershow AG, Lewis B, Treat-Jacobson DJ, Walsh ME, Oldenburg N, Regensteiner JG; CLEVER Research Group. Design of the multicenter standardized supervised exercise training intervention for the claudication: exercise vs endoluminal revascularization (CLEVER) study. Vasc Med. 2009 Nov;14(4):313-21. doi: 10.1177/1358863X09102295. PMID 19808716
- [Background] Murphy TP, Hirsch AT, Cutlip DE, Regensteiner JG, Comerota AJ, Mohler E, Cohen DJ, Massaro J; CLEVER Investigators. Claudication: exercise vs endoluminal revascularization (CLEVER) study update. J Vasc Surg. 2009 Oct;50(4):942-945.e2. doi: 10.1016/j.jvs.2009.04.076. Epub 2009 Aug 5. PMID 19660897
- [Result] Murphy TP, Cutlip DE, Regensteiner JG, Mohler ER, Cohen DJ, Reynolds MR, Massaro JM, Lewis BA, Cerezo J, Oldenburg NC, Thum CC, Goldberg S, Jaff MR, Steffes MW, Comerota AJ, Ehrman J, Treat-Jacobson D, Walsh ME, Collins T, Badenhop DT, Bronas U, Hirsch AT; CLEVER Study Investigators. Supervised exercise versus primary stenting for claudication resulting from aortoiliac peripheral artery disease: six-month outcomes from the claudication: exercise versus endoluminal revascularization (CLEVER) study. Circulation. 2012 Jan 3;125(1):130-9. doi: 10.1161/CIRCULATIONAHA.111.075770. Epub 2011 Nov 16. PMID 22090168
- [Derived] Reynolds MR, Apruzzese P, Galper BZ, Murphy TP, Hirsch AT, Cutlip DE, Mohler ER 3rd, Regensteiner JG, Cohen DJ. Cost-effectiveness of supervised exercise, stenting, and optimal medical care for claudication: results from the Claudication: Exercise Versus Endoluminal Revascularization (CLEVER) trial. J Am Heart Assoc. 2014 Nov 11;3(6):e001233. doi: 10.1161/JAHA.114.001233. PMID 25389284